CLINICAL TRIAL: NCT02843282
Title: Brain & Cognitive Changes After Reasoning Training in Individuals With Bipolar Disorder
Brief Title: Reasoning Training in Individuals With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-16
Record Dates: First submitted 2016-07-14; First posted 2016-07-25 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Disorder; Cognitive Ability, General
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive training (Experimental): Advanced reasoning training
  Interventions: Behavioral: Advanced Reasoning Training

INTERVENTIONS:
Behavioral: Advanced Reasoning Training — This is a strategy-based intervention to enhance frontal lobe function. Strategies equip participants to improve their strategic attention, integrated reasoning, and innovation abilities.
  Other Names: Gist Reasoning Training

SUMMARY:
The purpose of this study is to examine cognitive and brain changes in individuals with bipolar disorder as a result of a cognitive training intervention.

DETAILED DESCRIPTION:
Participants will only include people who are fluent speakers of English, as not all of the standardized and experimental cognitive tests have been normed for non-English speakers. Participants will be screened for significant medical, neurological, or psychiatric illness other than bipolar disorder.

Participants will complete baseline cognitive testing. Reasoning training will take place in small groups, once a week for 2hr/session. After the training, participants will complete the cognitive testing again. A subset of participants who qualify for the brain imaging component will also complete a pre-post resting state brain scan.

Training effects will be measured behaviorally in trained areas (reasoning & physical) and untrained cognitive areas. Additionally, structural and functional brain imaging will measure changes in cerebral blood flow, global and regional brain volume, white matter tracts, efficiency, activation patterns, and blood oxygenation with a particular focus on changes to frontal regions.

Screening Session: A research assistant will conduct screening procedures over the phone including a brief medical questionnaire covering their history, current medications and any pre-existing conditions. Prior diagnosis of bipolar disorder and euthymic state will be confirmed with participant's psychiatrist or treating physician.

Neurocognitive Testing Session: A clinician will administer a group of standardized and experimental tests to each participant for each of the cognitive testing sessions. This session may last up to 3 hours, depending on the pace of the participant's response times. The intent of the tasks is to assess higher level thinking skills, working memory, and selective learning.

Functional magnetic resonance imaging (fMRI): Participants will have fMRI, at each aforementioned time point in the study, during which they will lie in the scanner while images of their brain will be recorded. Each session will take up to 90 minutes. During the fMRI and during the diffusion tensor imaging (DTI) the patient will be asked just to lie still.

Cognitive reasoning training: The gist-based reasoning training will be delivered in one, two hour session each week over 4 weeks. It is strategy-based rather than content-based so that the focus is not content specific or situation-dependent. Gist-based reasoning has been linked to frontal lobe activation and to measures of executive function.

Post Intervention: Following the intervention, patients will repeat the cognitive neuropsychological assessment and fMRI identical to the pre-training assessment. Participants are not paid for any of these tests or training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Must have physician or psychiatrist authorization form confirming participant fulfills 4 criteria:

  1. has diagnosis of Bipolar I or II
  2. has been stable and consistent with medication for last 3 months
  3. is in a euthymic, rather than manic or depressive, state
  4. is appropriate for a group-based intervention

     EXCLUSION CRITERIA:
* Not a native English speaker
* Less than 12 years education
* Additional psychiatric diagnosis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, PhD, Principal Investigator — The University of Texas at Dallas

IPD SHARING:
Plan to Share IPD: No
Not at this time

REFERENCES:
- [Background] Demant KM, Vinberg M, Kessing LV, Miskowiak KW. Effects of Short-Term Cognitive Remediation on Cognitive Dysfunction in Partially or Fully Remitted Individuals with Bipolar Disorder: Results of a Randomised Controlled Trial. PLoS One. 2015 Jun 12;10(6):e0127955. doi: 10.1371/journal.pone.0127955. eCollection 2015. PMID 26070195
- [Background] Preiss M, Shatil E, Cermakova R, Cimermanova D, Ram I. Personalized cognitive training in unipolar and bipolar disorder: a study of cognitive functioning. Front Hum Neurosci. 2013 May 13;7:108. doi: 10.3389/fnhum.2013.00108. eCollection 2013. PMID 23717272
- [Background] Deckersbach T, Nierenberg AA, Kessler R, Lund HG, Ametrano RM, Sachs G, Rauch SL, Dougherty D. RESEARCH: Cognitive rehabilitation for bipolar disorder: An open trial for employed patients with residual depressive symptoms. CNS Neurosci Ther. 2010 Oct;16(5):298-307. doi: 10.1111/j.1755-5949.2009.00110.x. PMID 19895584
- [Background] Chapman SB, Mudar RA. Enhancement of cognitive and neural functions through complex reasoning training: evidence from normal and clinical populations. Front Syst Neurosci. 2014 Apr 28;8:69. doi: 10.3389/fnsys.2014.00069. eCollection 2014. PMID 24808834
- [Derived] Venza EE, Chapman SB, Aslan S, Zientz JE, Tyler DL, Spence JS. Enhancing Executive Function and Neural Health in Bipolar Disorder through Reasoning Training. Front Psychol. 2016 Nov 1;7:1676. doi: 10.3389/fpsyg.2016.01676. eCollection 2016. PMID 27847486

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled participants were excluded from the training
Period: Overall Study
Arm/Group | Cognitive Training
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All baseline participants completed study.
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline: Test of Strategic Learning
Description: Complex abstraction subtest: After reading a complex text, participants generate a high-level synthesis of abstracted ideas (versus recall of concrete details). [raw scores, min value = 0, max value = 10, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 2.35 (0.32)
  post | 3.04 (0.32)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.040, Regression, Linear; Mean Difference (Net) = 0.69

2. Secondary Outcome: Change From Baseline: Wechsler Adult Intelligence Scale (WAIS), Similarities Subtest
Description: Participants are provided with two words/concepts and must state how they are alike; [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 12.63 (0.40)
  post | 13.62 (0.41)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.004, Regression, Linear; Mean Difference (Net) = 0.98

3. Secondary Outcome: Change From Baseline: Delis-Kaplan Executive Function System (DKEFS) Card Sorting
Description: Participants must sort a set of cards into as many groups as possible, based on certain parameters. This score reflects the correct number of sorts generated. [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.70 (0.42)
  post | 13.56 (0.42)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = 1.95

4. Secondary Outcome: Change From Baseline: Working Memory (Digits Backwards)
Description: Participants must recite number sequences in reverse order; [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 6.78 (0.36)
  post | 7.30 (0.36)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.039, Regression, Linear; Mean Difference (Net) = 0.52

5. Secondary Outcome: Change From Baseline: Delis-Kaplan Executive Function System (DKEFS) Color-Word, Inhibition & Switching Subtest
Description: Participants must either state color of word or read the word presented; [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.04 (0.37)
  post | 11.46 (0.37)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.092, Regression, Linear; Mean Difference (Net) = 0.42

6. Secondary Outcome: Change From Baseline: Divided Attention
Description: Participants connect letters and numbers in ascending order as quickly as they can; [raw score in seconds, min value = 0, max value = 200, lower indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
seconds
  pre | 73.44 (5.43)
  post | 66.86 (5.48)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.052, Regression, Linear; Mean Difference (Net) = 6.58

7. Secondary Outcome: Change From Baseline: Verbal Fluency
Description: Participants had to generate as many words as possible in one minute that fit task parameters; [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.30 (0.61)
  post | 11.82 (0.61)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.121, Regression, Linear; Mean Difference (Net) = 0.52

8. Secondary Outcome: Change From Baseline: Rey Auditory Verbal Learning Test (RAVLT)
Description: Participants are asked to recall a list of words they heard 20 minutes earlier; [raw scores, min value = 0, max value = 15, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 9.70 (0.68)
  post | 10.93 (0.68)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.019, Regression, Linear; Mean Difference (Net) = 1.23

9. Secondary Outcome: Change From Baseline: Logical Memory
Description: Participants are asked to recall the details of a story they were read 20 minutes earlier; [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.89 (0.72)
  post | 12.26 (0.72)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.278, Regression, Linear; Mean Difference (Net) = 0.37

10. Secondary Outcome: Change From Baseline: Quality of Life in Bipolar Disorder (QoL.BD)
Description: Participants fill out a self-report questionnaire assessing different domains of quality of life; [raw score; min value = 0, max value = 280, higher score indicates higher reported quality of life]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 176.93 (6.90)
  post | 183.93 (7.00)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.095, Regression, Linear; Mean Difference (Net) = 7

11. Secondary Outcome: Resting State Relative Cerebral Brain Blood Flow (rCBF)
Description: Mean-level change in resting state relative cerebral brain blood flow (rCBF) in left Inferior frontal gyrus (min value = 0, max value = 2, lower value indicates decreased cerebral blood flow and higher indicates increased cerebral blood flow)
Time Frame: Pre (from baseline) and within 2 weeks post intervention
Population: Only for participants who participated in brain imaging portion of study (only for participants that were eligible for MRI)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 12
score on a scale
  pre | 0.67 (0.11)
  post | 0.82 (0.10)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Other; p < 0.01, Whole brain voxel-wise correlation analy; Mean Difference (Net) = 0.15

12. Secondary Outcome: Change From Baseline: Delis-Kaplan Executive Function System (DKEFS) Accurate Description of Sorts
Description: Participants must sort a set of cards into as many groups as possible, based on certain parameters, and state why it is an accurate sort. This score reflects the accuracy of the sort description. [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.74 (0.43)
  post | 12.96 (0.43)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.001, Regression, Linear; Mean Difference (Net) = 1.22

13. Secondary Outcome: Change From Baseline: Delis-Kaplan Executive Function System (DKEFS) Accurate Recognition of Sorts
Description: After proctor has sorted cards, participants must state why sort is accurate/how cards are alike. [scaled scores, min value = 0, max value = 19, higher indicates better performance]
Time Frame: Pre and within 2 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Training
Number analyzed (Participants) | 27
score on a scale
  pre | 11.56 (0.47)
  post | 12.89 (0.47)
Statistical Analysis 1: Comparison: Cognitive Training; Test type: Superiority; p = 0.007, Regression, Linear; Mean Difference (Net) = 1.33

ADVERSE EVENTS:
Time Frame: Baseline assessment to post assessment (2 weeks post intervention)
Arm/Group | Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT02843282/Prot_SAP_ICF_000.pdf